CLINICAL TRIAL: NCT03858842
Title: Non-interventional Study Describing Epidemiology, Clinical Characteristics, Prognosis and Healthcare Costs of PF-ILD and SSc-ILD Patients in France, 2010-2017
Brief Title: Non-interventional Study Describing Epidemiology, Prognosis and Patient Healthcare Costs in France, 2010-2017
Acronym: PROGRESS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0027
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-02

CONDITIONS: Lung Diseases, Interstitial; Lung Disease With Systemic Sclerosis
Keywords: Progressive fibrosing interstitial lung disease; Systemic Sclerosis-Associated Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Health Care Costs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PF-ILD and SSc-ILD patients: PF-ILD and SSc-ILD patients
  Interventions: Other: epidemiology, healthcare costs in non-IPF PF-ILD and SSc-ILD

INTERVENTIONS:
Other: epidemiology, healthcare costs in non-IPF PF-ILD and SSc-ILD — epidemiology, characteristics, healthcare resources and associated costs of patients diagnosed with non-IPF PF-ILD and SSc-ILD

SUMMARY:
Interstitial lung diseases (ILDs) are a heterogeneous group of disorders, which encompass a wide range of conditions. In some patients with fibrosing ILDs, a progressive phenotype similar to that observed in idiopathic pulmonary fibrosis (IPF) may develop during the course of the disease (PF-ILD), including patients with systemic sclerosis (SSc)-related ILD.

The aim of the study is to estimate the incidence and prevalence and to describe the characteristics of patients diagnosed with non-IPF PF-ILD and SSc-ILD, to describe the natural course of disease, and to explore the correlation between mortality and Forced Vital Capacity (FVC) of the patients with non-IPF PF-ILD.

This study will be based on two data sources: the French national medico administrative database (SNDS) and the ILD cohort from the National French center for rare pulmonary diseases in Lyon, France.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for PF-ILD and SSc-ILD in France between 01/01/2010 and 31/12/2017
* Men or women aged ≥ 18 years old at diagnosis

Exclusion Criteria:

* Patients treated by anti-fibrotic
* Patients diagnosed with IPF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for SSc-ILD, and PF-ILD (excluding the IPF patients)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of PF-ILD and SSc-ILD patients | Between 2010 and 2017
  The study will describe for the non-idiopathic pulmonary fibrosis (IPF) progressive fibrosing interstitial lung (PF-ILD) and Systemic Sclerosis-Associated Interstitial Lung Disease (SSc-ILD) patients in France.:
  * the epidemiology (incidence and prevalence),
  * the characteristics of patients,
  * the healthcare resource use and associated costs
Prevalence of PF-ILD and SSc-ILD patients | Between 2010 and 2017
  The study will describe for the non-idiopathic pulmonary fibrosis (IPF) progressive fibrosing interstitial lung (PF-ILD) and Systemic Sclerosis-Associated Interstitial Lung Disease (SSc-ILD) patients in France.:
  * the epidemiology (incidence and prevalence),
  * the characteristics of patients,
  * the healthcare resource use and associated costs
characteristics of PF-ILD and SSc-ILD patients | Between 2010 and 2017
  The study will describe for the non-idiopathic pulmonary fibrosis (IPF) progressive fibrosing interstitial lung (PF-ILD) and Systemic Sclerosis-Associated Interstitial Lung Disease (SSc-ILD) patients in France.:
  * the epidemiology (incidence and prevalence),
  * the characteristics of patients,
  * the healthcare resource use and associated costs
healthcare resource use of PF-ILD and SSc-ILD patients | Between 2010 and 2017
  The study will describe for the non-idiopathic pulmonary fibrosis (IPF) progressive fibrosing interstitial lung (PF-ILD) and Systemic Sclerosis-Associated Interstitial Lung Disease (SSc-ILD) patients in France.:
  * the epidemiology (incidence and prevalence),
  * the characteristics of patients,
  * the healthcare resource use and associated costs
associated costs of PF-ILD and SSc-ILD patients | Between 2010 and 2017
  The study will describe for the non-idiopathic pulmonary fibrosis (IPF) progressive fibrosing interstitial lung (PF-ILD) and Systemic Sclerosis-Associated Interstitial Lung Disease (SSc-ILD) patients in France.:
  * the epidemiology (incidence and prevalence),
  * the characteristics of patients,
  * the healthcare resource use and associated costs

SECONDARY OUTCOMES:
mortality for the non-idiopathic pulmonary fibrosis (IPF) progressive fibrosing interstitial lung (PF-ILD) in France. | Between 2010 and 2017
  correlation between mortality and FVC for the non-idiopathic pulmonary fibrosis (IPF) progressive fibrosing interstitial lung (PF-ILD) in France.
Forced Vital Capacity for the non-idiopathic pulmonary fibrosis (IPF) progressive fibrosing interstitial lung (PF-ILD) in France. | Between 2010 and 2017
  correlation between mortality and FVC for the non-idiopathic pulmonary fibrosis (IPF) progressive fibrosing interstitial lung (PF-ILD) in France.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Cottin, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Cardiologique Louis Pradel, Bron, France

REFERENCES:
- [Derived] Cottin V, Larrieu S, Boussel L, Si-Mohamed S, Bazin F, Marque S, Massol J, Thivolet-Bejui F, Chalabreysse L, Maucort-Boulch D, Jouneau S, Hachulla E, Chollet J, Nasser M. Epidemiology, Mortality and Healthcare Resource Utilization Associated With Systemic Sclerosis-Associated Interstitial Lung Disease in France. Front Med (Lausanne). 2021 Aug 30;8:699532. doi: 10.3389/fmed.2021.699532. eCollection 2021. PMID 34552943
- [Derived] Nasser M, Larrieu S, Boussel L, Si-Mohamed S, Bazin F, Marque S, Massol J, Thivolet-Bejui F, Chalabreysse L, Maucort-Boulch D, Hachulla E, Jouneau S, Le Lay K, Cottin V. Estimates of epidemiology, mortality and disease burden associated with progressive fibrosing interstitial lung disease in France (the PROGRESS study). Respir Res. 2021 May 24;22(1):162. doi: 10.1186/s12931-021-01749-1. PMID 34030695
- [Derived] Nasser M, Larrieu S, Si-Mohamed S, Ahmad K, Boussel L, Brevet M, Chalabreysse L, Fabre C, Marque S, Revel D, Thivolet-Bejui F, Traclet J, Zeghmar S, Maucort-Boulch D, Cottin V. Progressive fibrosing interstitial lung disease: a clinical cohort (the PROGRESS study). Eur Respir J. 2021 Feb 11;57(2):2002718. doi: 10.1183/13993003.02718-2020. Print 2021 Feb. PMID 32943410